CLINICAL TRIAL: NCT05327062
Title: CRT-DRIVE: Cardiac Resynchronization Therapy Delivery Guided Non-Invasive Electrical and Venous Anatomy Assessment
Brief Title: Cardiac Resynchronization Therapy Delivery Guided Non-Invasive Electrical and Venous Anatomy Assessment
Acronym: CRT-DRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: XSpline S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRT-DRIVE_01
Record Dates: First submitted 2022-03-22; First posted 2022-04-14 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Resynchronization Therapy; Chronic Heart Failure; Left Bundle-Branch Block
Keywords: Non-invasive activation mapping; Coronary Sinus
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: The investigation will include 9 European and 4 US investigational sites. The goal is to enroll a total number of 150 patients. It is expected about 1.5 patients per site per month over a period of maximum 8 months after site opening. The study duration is set at 12-month, 6 months for patient enrollment and 6 months of follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CRT implantation guided by XSpline (Experimental): The sample size estimation was based on two recent studies including CRT patients with similar clinical and demographic characteristics as in this study: the SMART-MSP and the SMART CRT. The SMART-MSP is a prospective, observational study that enrolled 584 CRT recipients at 52 US sites. In a typical modern CRT population, 75% of patients had a reduction of the end-systolic volume ≥ 15% at 6-month follow-up. The SMART-CRT study enrolled 699 CRT patients randomized to a treatment arm and a control group. At 6-months follow-up, a reduction of LVESV ≥15% was achieved for 67.7% of the patients in the control group and for 74.8% of those in the treatment arm. Therefore, it is assumed that in a modern CRT population at least 70% of the patients will have a reduction of the LVESV ≥15% of the baseline value at 6-months after CRT implantation. To demonstrate that this proportion of patients can be equally achieved with the approach tested in this study at least 150 patients need to be included.
  Interventions: Device: CRT implantation guided by XSpline, a non-invasive electrical and venous anatomy assessment

INTERVENTIONS:
Device: CRT implantation guided by XSpline, a non-invasive electrical and venous anatomy assessment — The following information and data will be obtained from the routine clinical work up of the patients: Patient demographics, cardiovascular medical history, and clinical examination; 12-lead ECG; Standard echocardiography; Computed tomography angiography for visualization of atria, ventricle, and coronary sinus.
  Imaging data will be transferred to the cloud-based web-platform using a dedicated software provided by study sponsor. Data processing includes evaluating the quality of the data and calculation of various anatomical and electrical parameters, and identification of the target zone as a point in the target vein closest to the latest activation zone.
  LV-lead location is based on the information provided by the dedicated software followed by visual X-ray based verification of anatomically suitable/most desirable position.
  The patient will undergo CRT device implantation according to local protocols.

SUMMARY:
The objective of this prospective, multicenter controlled study is to assess the feasibility of a patient-tailored implantation by creating a cloud-based pre-procedural multimodality CRT-roadmap by integration of 3D images from 3D activation sequence from ECG, and coronary venous anatomy from cardiac computed tomography. This CRT-roadmap will be used to guide LV lead placement to a coronary vein in an electrically late-activated region.

Study Hypothesis: At least 75% of patients undergoing a CRT implantation guided by non-invasive electrical and venous anatomy assessment (XSPLINE technology) will show a reduction of left ventricular end-systolic volume of 15% or more at 6-month evaluation.

ELIGIBILITY:
Eligible subjects shall meet all following criteria:

* Appropriately signed and dated informed consent.
* Age ≥18 years at time of consent.
* CRT indication according to the 2021 ESC guidelines on cardiac pacing and CRT (class I and IIA indication in patients with LBBB QRS morphology) or to 2017 AHA/ACC/HFSA guidelines (COR I).
* Sinus rhythm
* QRS duration ≥130 ms
* Left bundle branch block
* Left ventricular ejection fraction ≤35%
* Symptomatic heart failure NYHA class ≥ II
* Documented stable medical treatment for at least 6 months
* No cardiovascular intervention during the last 6 month

Exclusion Criteria are:

* History of persistent or permanent atrial fibrillation
* Previous pacemaker or ICD implantation
* Indication to pacing due to bradycardia
* Patients considered for His bundle pacing or cardiac conduction pacing
* Patients with unstable angina
* Subject experienced a recent myocardial infarction, within 40 days prior to enrollment
* Subject underwent coronary artery bypass graft or valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation, or is actively listed on the transplantation list, or has reasonable probability (per investigator's discretion) of undergoing transplantation in the next year
* Subject is implanted with a left ventricular assist device
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure
* Subject has severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated within study period)
* Subject has congenital heart disease
* Subject has a mechanical right-sided heart valve
* Subject has a life expectancy of less than one year in the opinion of the investigator
* Pregnant or breastfeeding women, or women of child bearing potential and who are not on a reliable form of birth control
* Subject is enrolled in one or more concurrent studies that would confound the results of this study
* Patients who have contraindications to CT scanning.
* Patients with chronic kidney diseases and estimated glomerular filtration rate (eGMR) calculated based on CKD-EPI 2009 < 40 ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Reduction of left ventricular end-systolic volume of at least 15% in 75% of CRT treated patients | 6 months follow-up
  Increase in efficacy of CRT using XSpline technology assessed by reduction of left ventricular end-systolic volume of at least 15% at 6-month follow-up in 75% of CRT treated patients, based on routine echo-cardiographic measurements

SECONDARY OUTCOMES:
Feasibility of systematic use of XSpline platform for CRT implantation | 6 months follow-up
  Feasibility of systematic use of automatic cloud-based, AI-based XSpline technology through statistics on software performance (e.g. percentage of core tasks completed higher than defined thresholds)
CRT procedural time difference | 6 months follow-up
  Evaluate the change in CRT procedural time by comparing with standard approach as found in literature, time in minutes
Total X-ray exposure time difference | 6 months follow-up
  Evaluate the change in total X-ray exposure time by comparing with standard approach as found in literature, time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Auricchio, MD PhD FESC, Principal Investigator — Istituto Cardiocentro Ticino
Locations (13):
- United States (4):
  - Rush University Medical center, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University Hospital, Durham, North Carolina
- Ordensklinikum Linz Elisabethinen Hospital, Linz, Austria
- Semmelweis University, Budapest, Hungary
- Italy (4):
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia
  - University Tor Vergata, Roma, Roma
  - General Hospital of Bolzano, Bolzano
  - Ospedale S. Maria del Carmine di Rovereto, Rovereto
- Maastricht University Medical Center, Maastricht, Netherlands
- Univeristat de Barcelona, Barcelona, Spain
- Istituto Cardiocentro Ticino, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Andrassy KM. Comments on 'KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease'. Kidney Int. 2013 Sep;84(3):622-3. doi: 10.1038/ki.2013.243. No abstract available. PMID 23989362
- [Background] Ramanathan C, Ghanem RN, Jia P, Ryu K, Rudy Y. Noninvasive electrocardiographic imaging for cardiac electrophysiology and arrhythmia. Nat Med. 2004 Apr;10(4):422-8. doi: 10.1038/nm1011. Epub 2004 Mar 14. PMID 15034569
- [Background] Cluitmans MJ, Peeters RL, Westra RL, Volders PG. Noninvasive reconstruction of cardiac electrical activity: update on current methods, applications and challenges. Neth Heart J. 2015 Jun;23(6):301-11. doi: 10.1007/s12471-015-0690-9. PMID 25896779
- [Background] Pezzuto S, Prinzen FW, Potse M, Maffessanti F, Regoli F, Caputo ML, Conte G, Krause R, Auricchio A. Reconstruction of three-dimensional biventricular activation based on the 12-lead electrocardiogram via patient-specific modelling. Europace. 2021 Apr 6;23(4):640-647. doi: 10.1093/europace/euaa330. PMID 33241411
- [Background] Zubarev S, Chmelevsky M, Budanova M, Trukshina M, Lyubimtseva T, Lebedeva V, et al. Non-invasive electrophysiological mapping in assessment of association of cardiac resynchronization effect from position of left ventricular electrode. Europace 2017;19(suppl_3):iii326-iii326. doi: 10.1093/ehjci/eux158.182
- [Background] Zubarev S, Chmelevsky M, Budanova M, Ryzhkov AV, Trukshina M, Lebedeva V, et al. Comparison of the late activation zone and the changes in the structure of the left ventricular myocardium in candidates for cardiac resynchronization therapy. Europace 2018;20(suppl_1):i54-i54. doi: 10.1093/europace/euy015.145
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822